CLINICAL TRIAL: NCT00851305
Title: Comparison Confocal Laser Endomicroscopy With Conventional Endoscopy for the Detection of Early Gastric Cancers
Brief Title: Detection of Early Gastric Cancers Using Confocal Laser Endomicroscopy
Acronym: CLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Chief of the Department of Gastroenterology, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008SDU-QILU-G01; 2006GG3202022; 2007(Ministry of Health)
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Stomach Neoplasms; Precancerous Conditions
Keywords: Stomach; endoscopy; neoplasms
MeSH Terms: conditions — Stomach Neoplasms; Precancerous Conditions; Neoplasms | interventions — Gastroscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 confocal laser endomicroscopy (Experimental): Targeted biopsies are performed when the lesion was considered as IM, dysplasia or carcinoma by confocal laser endomicroscopy.
  Interventions: Device: Endomicroscope (Pentax, Tokyo, Japan)
- 2 Conventional endoscopy (Active Comparator): Routine biopsies are performed when the lesion was considered as IM, dysplasia or carcinoma by conventional endoscopy.
  Interventions: Device: Gastroscopes (Pentax, Tokyo, Japan)

INTERVENTIONS:
Device: Endomicroscope (Pentax, Tokyo, Japan) — A Pentax EC3870K endomicroscope which can produce conventional white light endoscopic images and confocal images at the same time with a optical slice thickness of 7 μm, a lateral resolution of 0.7 μm, a scanning depth of 0 to 250 μm, a pixel density of 1024×512 pixels (at an image acquisition rate of 1.6 frames/second)，and a field of view of 475 μm×475 μm.
  Other Names: Pentax EC3870K endomicroscope
  Arms: 1 confocal laser endomicroscopy
Device: Gastroscopes (Pentax, Tokyo, Japan) — Conventional white light gastroscopes (Pentax EG-2940 gastroscopes)
  Other Names: Pentax EG-2940 gastroscopes (Pentax, Tokyo, Japan)
  Arms: 2 Conventional endoscopy

SUMMARY:
The purpose of this study is to determine whether endomicroscopy can improve the detection of Early Gastric Cancers (EGC).

DETAILED DESCRIPTION:
Endoscopy is proved to be the best method to achieve early diagnosis of gastric cancer (GC). Confocal laser endomicroscopy (CLE), a new diagnostic modality, has been shown to be valuable in increasing the diagnostic yield of colorectal neoplasias, but it is not clear whether CLE is helpful to find out early gastric cancer (EGC).The aim of the study is to investigate the value of CLE in improving the detection of EGCs.

ELIGIBILITY:
Inclusion Criteria:

* 45 years old ≤ age < 80 years old
* Patients with dyspeptic symptoms or with gastric premalignant conditions for surveillance gastroscopy

Exclusion Criteria:

* Known cancers or gastrectomy
* Scheduled for endoscopic treatment
* Alarm symptoms such as dysphagia, anaemia, gastrointestinal bleeding or obstruction, marked weight loss
* Under conditions such as:

  * ascites
  * jaundice
  * liver cirrhosis
  * impaired renal function
  * coagulopathy
  * fever
  * pregnancy
  * breastfeeding
* Inability to provide informed consent
* Known allergy to fluorescein sodium

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1786 (Actual)
Dates: Start 2008-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To compare the rate of EGCs/GCs using CLE versus conventional gastroscopy. | one year

SECONDARY OUTCOMES:
To evaluate the efficacy of in vivo CLE on different pathological characteristics of EGCs. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD. MD., Study Director — Department of Gastroenterology, Qilu Hospital, Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China